CLINICAL TRIAL: NCT02231216
Title: The Role of Turbinectomy in Rhinoseptoplasty: a Randomized Clinical Trial With Evaluation of Quality of Life
Brief Title: Quality of Life Study About the Role of Turbinectomy in Rhinoseptoplasty
Acronym: WHOQOL-BREF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 130516
Record Dates: First submitted 2014-09-02; First posted 2014-09-04 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Deviated Nasal Septum; Nasal Septal Defect; Nasal Septum, Irregular
Keywords: rhinoseptoplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rhinoseptoplasty and turbinectomy (Experimental): Patients submitted to rhinoseptoplasty associated to Endoscopic partial turbinectomy.
  Interventions: Procedure: Rhinoseptoplasty; Procedure: Partial turbinectomy; Procedure: Endoscopic partial turbinectomy
- Rhinoseptoplasty (Active Comparator): Patients submitted only to rhinoseptoplasty, without turbinectomy procedure.
  Interventions: Procedure: Rhinoseptoplasty

INTERVENTIONS:
Procedure: Rhinoseptoplasty — Rhinoseptoplasty without turbinectomy procedure
Procedure: Partial turbinectomy — After medial dislocation of the inferior turbinate, proceed partial resection of the inferior turbinate in all its inferior extension in range. Possible bleeding is cauterized.
  Other Names: Turbinectomy
  Arms: Rhinoseptoplasty and turbinectomy
Procedure: Endoscopic partial turbinectomy — Endoscopy to medial dislocation of the inferior turbinate with instrument
  Arms: Rhinoseptoplasty and turbinectomy

SUMMARY:
Research Question: Performing partial turbinectomy associated with rhinoseptoplasty is responsible for an increase in quality of life related to nasal obstruction when compared to no intervention in rhinoseptoplasty inferior turbinate?

* Population: patients eligible for functional rhinoseptoplasty and / or aesthetic
* Intervention: surgery, turbinectomy of inferior turbinates
* Comparison: the absence of intervention in inferior turbinates
* Primary endpoint: Quality of life related to nasal obstruction

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients to rhinoseptoplasty
* Patients who agreed to participate

Exclusion Criteria:

* Presence of symptoms of nasal obstruction in the absence of septal deviation, poor support of the nasal tip or clamping of the nasal valve;
* Presence of hypertrophic and obstructive inferior turbinates;
* Presence of sinonasal tumors;
* Patients undergoing treatment of other concomitant rhinoplasty entities such as inflammatory sinus pathology, adenoid hypertrophy, septal perforation, otoplasty and blepharoplasty.

Ages: 6 Months to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Quality of life related to nasal obstruction | 3 months
  Quality of life will be evaluated by the WHOQOL-BREF instrument, that comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment.

SECONDARY OUTCOMES:
Nasal sneezing | 3 MONTHS
  At 90 posoperative day patients were asked if they had nasal sneezing for more than one hour a day on most days, or not.
Nasal Rhinorrhea | 3 MONTHS
  At 90 posoperative day patients were asked if they had nasal rhinorrhea for more than one hour a day on most days, or not.
Nasal Pruritis | 3 MONTHS
  At 90 posoperative day patients were asked if they had nasal pruritis for more than one hour a day on most days, or not.
Allergic Conjunctivitis | 3 months
  At 90 posoperative day patients were asked if they had allergic conjunctivitis for more than one hour a day on most days, or not.
Topical Nasal Corticosteroids | 3 MONTHS
  At 90 posoperative day patients were asked if they were using topic nasal corticosteroids or not
Oral antihistamine | 3 months
  At 90 posoperative day patients were asked if they had used oral antihistamine in the past 30 days or not

CONTACTS AND LOCATIONS:
Overall Officials: Bianca H Moura, MD, Principal Investigator — Hospital de Clínicas de Porto Alegre; Michelle Lavinsky, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Garcia JPT, Moura BH, Rodrigues VH, Vivan MA, Azevedo SM, Dolci JEL, Migliavacca R, Lavinsky-Wolff M. Inferior Turbinate Reduction during Rhinoplasty: Is There Any Effect on Rhinitis Symptoms? Int Arch Otorhinolaryngol. 2021 Aug 5;26(1):e111-e118. doi: 10.1055/s-0041-1726046. eCollection 2022 Jan. PMID 35096167
- [Derived] de Moura BH, Migliavacca RO, Lima RK, Dolci JEL, Becker M, Feijo C, Brauwers E, Lavinsky-Wolff M. Partial inferior turbinectomy in rhinoseptoplasty has no effect in quality-of-life outcomes: A randomized clinical trial. Laryngoscope. 2018 Jan;128(1):57-63. doi: 10.1002/lary.26831. Epub 2017 Aug 16. PMID 28815717